CLINICAL TRIAL: NCT03934151
Title: Multicenter National Observational Study on Intracorporeal Versus Extracorporeal Technique for Ileocolic Anastomosis in Laparoscopic Right Hemicolectomy
Brief Title: Intracorporeal Versus Extracorporeal Technique for Ileocolic Anastomosis in Laparoscopic Right Hemicolectomy
Acronym: CoDIG
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gabriele Anania, Professore Associato, University Hospital of Ferrara
Other Study IDs: 170595
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-02

CONDITIONS: Complication of Gastrointestinal Anastomosis; Intestinal Anastomosis Complication
Keywords: laparoscopy; ileocolic anastomosis; right hemicolectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intracorporeal anastomosis: patients who underwent elective right hemicolectomy whose ileocolic anastomosis was performed with intracorporeal technique
  Interventions: Procedure: intracorporeal ileocolic anastomosis
- extracorporeal anastomosis: patients who underwent elective right hemicolectomy whose ileocolic anastomosis was performed with extracorporeal technique
  Interventions: Procedure: extracorporeal ileocolic anastomosis

INTERVENTIONS:
Procedure: intracorporeal ileocolic anastomosis — laparoscopic bowel transection and ileocolic anastomosis performed inside the abdomen with specimen retrieval in plastic bag
  Groups: intracorporeal anastomosis
Procedure: extracorporeal ileocolic anastomosis — ileocolic anastomosis is carried out by exteriorizing the bowel through a limited laparotomy
  Groups: extracorporeal anastomosis

SUMMARY:
The aim of the study is to analyze the postoperative complication rate of intracorporeal versus extracorporeal anastomotic technique in laparoscopic or video assisted right hemicolectomy for malignant and benign neoplasms . The lead center is the General and Thoracic Surgery Department of the University of Ferrara. Prof. Anania is the responsible for the enrollment of patients and the coordination with the collaborating centers in the six month-study

DETAILED DESCRIPTION:
CoDIG is a cohort, observational, prospective, multi-centric national study about ileo-colic anastomosis performing with EC or IC Technique during right laparoscopic hemicolectomy.

The observational period lasts from march 2018 and September 2018. The promoter of the study is "Istituto di Chirurgia Generale 1" of Ferrara University Hospital.

135 Italian Hospitals, accredited by Health Ministry, have been contacted via e-mail and all data was compiled into a web accessible SICE database, 85 Italian clinical centres, with demonstrated experience in colorectal laparoscopic surgery, have joined the study.

Every centre was asked not to change its surgical habits concerning the technologies used, the surgical approach, the anastomotic method, the post-operative management.

Every patient involved into the study was asked to sign a consent form in order to the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* Patients and/or legal guardians exhaustively informed by the investigator, and who have voluntarily provided written informed consent or, when unable to read and/or write, verbal consent put into writing by a third person
* Patients who underwent elective laparoscopic or video assisted right hemicolectomy at U.O. General and Thoracic Surgery for malignant or bening pathology.
* Patients who had prior chemotherapy and radiotherapy

Exclusion Criteria:

* Patients operated in emergency
* Pregnant women
* Right laparotomic hemicolectomy
* BMI> 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by malignant or benign pathology of the right colon treated in italian surgical centers accredited by the Ministry of Public Health
Sampling Method: Non-Probability Sample
Enrollment: 1225 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Anastomotic complications | maximum 30 days
  number of anastomotic complications after right hemicolectomy when ileocolic anastomosis is performed with intracorporeal or extracorporeal technique
Postoperative day of discharge | 4 to 30 days
  the lenght of stay in hospital measured in days after right hemicolectomy with ileocolic anastomosis performed with intracorporeal or extracorporeal technique

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Anania, Principal Investigator — Società Italiana Chirurgia Endoscopica
Locations (85):
- Italy (85):
  - ULSS5 Polesa - Ospedale di Adria, Adria
  - San Lazzaro Alba, Alba
  - Ospedale Civile L. Bonomo, Andria
  - "U.Parini" di AOsta, Aosta
  - Ospedale C e G Mazzoni, Ascoli Piceno
  - Casa di Cura Villa Maria, Avellino
  - Ospedale di Bassano del Grappa, Bassano del Grappa
  - Policlinico San Marco, Bergamo
  - Ospedale Maggiore di Bologna, Bologna
  - SS. Pietro e Paolo, Borgosesia
  - ASST Spedali Civili, Brescia
  - Spedali Civili di Brescia Presidio Montichiari, Brescia
  - Policlinico Universitario di Monserrato - AOU Cagliari, Cagliari
  - Santissima Trinità, Cagliari
  - Aslto5 Piemonte, Chieri
  - Bassini, Cinisello Balsamo
  - U.O. Chirurgia Cles, Cles
  - Santa Maria dei Battuti, Conegliano
  - Aso Santa Croce E Carle Di Cuneo, Cuneo
  - Regina Montis Regalis Mondovì, Cuneo
  - Ospedale "E. Profili" Fabriano, Fabriano
  - Arcispedale Sant'Anna Ferrara, Ferrara
  - Istituto di chirurgia generale 1, Ferrara
  - Ospedale di Fidenza; AUSL Parma, Fidenza
  - AOU Careggi, Florence
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Chirurgia d' Urgenza Careggi, Florence
  - Ospedali Riuniti di Foggia, Foggia
  - Ospedale Morgagni-Pierantoni, Forlì
  - Ospedale Policlinico San Martino, Genova
  - Chirurgia Gorizia, Gorizia
  - Gualdo Tadino, Gubbio
  - Carlo Urbani, Jesi,, Iesi
  - Ospedale Sant'Andrea, La Spezia
  - Ospedale Del Delta, Lagosanto
  - N.S. della Mercede, Lanusei
  - ICOT, Latina
  - AAS 2 "Bassa Friulana-Isontina", Ospedale di Latisana-Palmanova, Latisana
  - Ospedale Civile San Salvatore, L’Aquila
  - Policlinico G. Martino, Messina
  - "ASST NORD MILANO Ospedale Città di Sesto San Giovanni ", Milan
  - "ASST OVEST MILANESE - Ospedale G. Fornaroli Magenta ", Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IEO (Istituto Europeo di Oncologia), Milan
  - IRCCS Policlinico Ospedale Maggiore Milano, Milan
  - Ospedale Sacco, Milan
  - San Paolo, Milan
  - San Raffaele, Milan
  - OCSAE, Modena
  - Policlinico di Modena, Modena
  - San Valentino, Montebelluna
  - A.O.U. Federico II, Napoli
  - Int Pascale Napoli, Napoli
  - Monaldi, AORN, Napoli
  - San Francesco, Nuoro
  - Giovanni Paolo II, Olbia
  - San Luigi Gonzaga, Orbassano
  - Aoup P. Giaccone, Palermo
  - Città di Castello, Perugia
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ospedale civile, Pescara
  - Pederzoli, Peschiera del Garda
  - Ospedale Santa Corona, Pietra Ligure
  - Ospedale San Jacopo, Pistoia
  - Azienda Ospedaliera S. Maria degli Angeli, Pordenone
  - Ospedale San Tommaso dei Battuti- ULSS 4 Veneto orientale, Portogruaro
  - Santa Maria delle Croci, Ravenna
  - Chirurgia Generale, Riccione
  - Infermi, Rimini
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Azienda Ospedaliera Universitaria Policlinico "Umberto I", Roma
  - Ospedale San Camillo - Forlanini, Roma
  - ospedale San Filippo Neri Roma, Roma
  - Sant'Eugenio- Asl Roma2, Roma
  - Azienda Ospedaliera Universitaria " San Giovanni di Dio e Ruggi d'Aragona" - Università di Salerno, Salerno
  - Ospedale Nostra Signora di Bonaria, San Gavino Monreale
  - "A.O.U. Sassari ", Sassari
  - Ospedale Sassuolo SPA, Sassuolo
  - Policlinico Le Scotte, Siena
  - S. Vincenzo, Taormina
  - Citta della Salute e della Scienza di Torino sede Molinette, Torino
  - Cardinale Panico, Tricase
  - Azienda Sanitaria Universitaria Integrata di Trieste - Ospedale di Cattinara, Trieste
  - Ospedale Santa Maria della Misericordia, Udine
  - Sant'Andrea, Vercelli

IPD SHARING:
Plan to Share IPD: No
privacy

REFERENCES:
- [Derived] Anania G, Agresta F, Artioli E, Rubino S, Resta G, Vettoretto N, Petz WL, Bergamini C, Arezzo A, Valpiani G, Morotti C, Silecchia G; SICE CoDIG (Colon Dx Italian Group). Laparoscopic right hemicolectomy: the SICE (Societa Italiana di Chirurgia Endoscopica e Nuove Tecnologie) network prospective trial on 1225 cases comparing intra corporeal versus extra corporeal ileo-colic side-to-side anastomosis. Surg Endosc. 2020 Nov;34(11):4788-4800. doi: 10.1007/s00464-019-07255-2. Epub 2019 Nov 18. PMID 31741153